CLINICAL TRIAL: NCT06021730
Title: Utilization and Utility of Patient After-Visit Instructions at a University Rheumatology Outpatient Clinic: Status and Randomized Prospective Pilot Intervention Study
Brief Title: Impact of After Visit Instructions on Patient Comprehension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22072004
Record Dates: First submitted 2023-08-21; First posted 2023-09-01 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: After Visit Instructions; Patient Education; Teach-Back Communication; Patient Comprehension
Keywords: After Visit Summary; Readability; REALM; A-REALM
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients received standard after visit procedure based on the provider
- Standardized After Visit Instructions Only (Experimental): The standardized after visit instructions (AVI) only group included patients receiving typed standardized AVI which included a text template that providers used to write customized AVI for the patient.
  Interventions: Behavioral: Standardized After Visit Instructions Only
- Standardized After Visit Instructions & Teach Back (Active Comparator): The standardized AVI & teach back (TB) group included standardized written AVI with the patient repeating to the provider which changes and future management had been agreed upon during the visit.
  Interventions: Behavioral: Standardized After Visit Instructions & Teach Back

INTERVENTIONS:
Behavioral: Standardized After Visit Instructions Only — The intervention took a standardized approach to after visit instructions which included a customizable template that would review patients conditions, changes in any medications, and any future labs, imaging, or referrals.
  Arms: Standardized After Visit Instructions Only
Behavioral: Standardized After Visit Instructions & Teach Back — This intervention included the Standardized After Visit Instructions and included teach back, a process by which patients restate in their own words their understanding of their condition, what was discussed in the visit, and what potential changes were made
  Arms: Standardized After Visit Instructions & Teach Back

SUMMARY:
This prospective study aims to analyze the influence of standardized after visit instructions (AVI) and teach back (TB) method on patients' understanding of health information. The study divided routine clinic patients into three groups: standard care, standardized AVI, and standardized AVI with TB. Patient health literacy, satisfaction, and AVI comprehension were gauged through surveys and post-visit follow-up calls. The investigators hypothesized that there would be an improvement in patient comprehension with the standardized AVI or TB when compared to controls.

DETAILED DESCRIPTION:
This study seeks to investigate the discharge practices of the Rheumatology clinic and analyze whether variations in these practices impact patient satisfaction, enhance their comprehension of their disease, and potentially influence the progression of their condition. Participants agreeing to take part in this study will be engaged for a duration of up to three (3) weeks, encompassing two study visits-one during their regular clinic appointment and another through a telephone study visit.

During the initial in-person visit, participants will complete a health literacy survey before their appointment and a satisfaction survey afterward. Approximately 1-2 weeks following the in-person visit, participants will receive a telephone call to respond to questions regarding their visit. More details of the study are outlined below.

Prior to commencing the study, participants will be asked to provide their consent by signing a form indicating their willingness to take part. The participants will then be randomly allocated to one of three study groups: the Control Group, the After Visit Instructions (AVI) Group, or the AVI with teach back (TB) group.

Throughout the course of the study, participants will engage in various activities. First, they will complete a health literacy form, designed to assess their familiarity with commonly used terms in rheumatology clinics. This will take place prior to the standard clinic visit and is expected to last around 5 minutes.

During the regular clinic visit, participants will follow different protocols based on their assigned group:

* Participants in the Control Group will experience their usual clinic visit.
* Those in the AVI Group will receive a personalized set of After Visit Instructions (AVI) that detail any changes in their care. This additional interaction is anticipated to last approximately 2 minutes.
* Individuals in the AVI with TB Group will be asked to explain, in their own words, the modifications made during their visit. This interaction is expected to take an extra 1 minute.

After the clinic visit, all participants will complete a satisfaction survey, assessing both the provider's performance and their contentment with the discharge process. This survey is estimated to take around 3 minutes to complete.

During the follow-up period, participants will receive a phone call 1-2 weeks after their clinic visit to respond to inquiries regarding their appointment experience and the discharge process. This telephone interview is anticipated to take around 10 minutes and aims to gather valuable insights.

Furthermore, foundational data will be extracted from participants' electronic medical records. This information will encompass details such as gender, date of birth, ethnicity, race, specific disease information, ongoing medications, and data from forms filled out before each visit that provide a comprehensive view of disease activity.

This study incorporates medical data from electronic medical records while ensuring confidentiality. Risks include potential loss of privacy, although safeguards are implemented. The study may extend the clinic visit by a maximum of 15 minutes, with no other anticipated risks.

Potential benefits include enhanced discharge practices, including standardized AVI templates and the "teach back" method, which could improve disease comprehension and management adherence. However, responses to interventions can vary, so outcomes cannot be pre-determined.

Participation in the control group offers no anticipated benefits. This study is not a treatment study, and the only alternative to participation is non-participation.

ELIGIBILITY:
Inclusion Criteria:

- Patients seen in the Rush University Medical Center Rheumatology Clinic

Exclusion Criteria:

* Tele-medicine visits
* English is not the primary language. This is due to inability of all providers to provide custom AVI due to language limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Patient Comprehension Survey | 1-2 weeks after initial visit
  This is a telephone survey that will assess patients comprehension of disease over three main categories: disease state, medication changes, and referral/imaging/lab requests. Each category will be measure concordance of the patients understanding with what was written in the note in the form of a percentage from 0% to 100%. A higher percentage means a better understanding of ones disease.

SECONDARY OUTCOMES:
Patient Satisfaction Survey | Will receive in email or in person immediately after initial visit
  Patient satisfaction will be assessed through a in person or email survey that will assess multiple elements of satisfaction. A higher score indicates a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Hassan, MD, Principal Investigator — Rush University Medical Center Associate Professor Rheumatology Department
Locations (1):
- Rush University Medical Center Division of Rheumatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT06021730/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT06021730/ICF_001.pdf